CLINICAL TRIAL: NCT04360954
Title: Evaluation of Commerical Antibody Tests for COVID-19
Brief Title: Evaluation of Antibody Tests for COVID-19
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 202004088
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: COVID; Coronavirus
Keywords: COVID; Coronavirus; Antibody test kit
MeSH Terms: conditions — Coronavirus Infections | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Plasma or serum.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Acute COVID infection: Active infection with positive RT-PCR
  Interventions: Diagnostic Test: Diagnostic test
- Convalescent COVID: Recent documented infection. Now asymptomatic and RT-PCR negative.
  Interventions: Diagnostic Test: Diagnostic test
- US Controls: Human samples pre-COVID.
  Interventions: Diagnostic Test: Diagnostic test
- LMIC Controls: Samples from LMIC pre-COVID.
  Interventions: Diagnostic Test: Diagnostic test

INTERVENTIONS:
Diagnostic Test: Diagnostic test — There is no intervention. This study will test deidentified archived biosamples.

SUMMARY:
The purpose of this study is to evaluate the sensitivity and specificity of several marketed commercial or prototype test kits for antibody to SARS-CoV-2. The focus will be on rapid-format, point-of-care antibody test kits that detect both IgM and IgG antibodies to recombinant viral proteins.

Note: No voluntary enrolment into this study will be conducted; all testing is to be conducted anonymously.

DETAILED DESCRIPTION:
Background

Molecular (RT-PCR) tests are currently the gold standard for diagnosis of COVID-19. They detect viral RNA and are a good marker for current infection and infectivity. However, these tests are expensive and in short supply. In advanced COVID-19 cases, virus concentration in the upper respiratory tract is often low, as the infection has spread to the lungs and viral RNA is sometimes undetectable by RT-PCR using nasal swaps. Antibody tests detect human antibodies to viral proteins in the blood or other body fluids. They could be useful for diagnosing current infections (slightly less sensitive than RT-PCR tests), and they remain positive after persons have recovered from the infection. Thus, antibody tests are expected to be useful for diagnosis of current infections, for verifying recent infections in persons who were not tested by RT-PCR when they were ill, and for documenting possible immunity to the virus. Antibody tests may be especially valuable for use in low and middle income countries that lack resources for widespread molecular testing for SARS-CoV-2 infection.

Anticipated test sensitivity and specificity. Manufacturer data for several antibody tests claim that more than 90% of persons with COVID-19 (clinical symptoms and positive molecular tests) have positive antibody test results for IgM and/or IgG. They also claim specificity in the range of 93-95% for samples from persons who have not been exposed to SARS-CoV-2.

Availability of antibody tests. In recent months, many antibody tests have been developed and marketed. The Foundation for Innovative New Diagnostics (FIND, closely linked to World Health Organization (WHO) and supported by a large grant from the United Kingdom government) in Geneva Switzerland reported that they had identified more than 70 such tests, and they shortlisted 27 tests for further evaluation. Of these, only one test produced in the USA (produced by Cellex) has received an emergency use authorization (EUA) from the US FDA, and no test has formal FDA approval. Antibody tests use different diagnostic platforms, but most tests use the SARS-CoV-2 S1protein, and a few tests also use the SARS-CoV-2 N protein. Few studies that independently evaluated the performance of these rapid antibody tests have been published to date in peer-reviewed journals. Therefore, more data are needed to evaluate the sensitivity, specificity, and value of these tests.

Methods

The Weil Lab research group at Washington University School of Medicine (WUSM) has extensive experience developing and evaluating rapid format diagnostic tests for infectious diseases. The group has special interest in infectious disease diagnostics that can be used in low and middle income countries and is used to work under challenging conditions after disease outbreaks. In this project, rapid-format antibody tests for SARS-CoV-2 will be evaluated and antibody test results will be compared with results of RT-PCR and metadata (age, gender, clinical symptoms, time after exposure when known).

Patient samples. Deidentified serum or plasma samples will be tested from patients who have been hospitalized and tested positive for COVID-19. Control samples from our serum bank (deidentified samples from healthy humans and samples from persons with parasitic diseases) will also be tested. The number of serum or plasma samples to be tested will be left open, but this will depend in part on the number of samples available and the availability of test kits. It is anticipated that approximately 500 samples will be tested initially, but more may be tested if that is necessary to achieve study objectives. The tests and research are for research only, and we will not report test results from individual patient samples to clinicians to support patient care.

Note: No voluntary enrolment into this study will be conducted; all testing is to be conducted anonymously.

Antibody test kits. Marketed commercial or prototype antibody detection kits will be obtained by donation or purchase. Tests to be evaluated are to be determined, but this will depend on availability and cost. The focus will be on rapid-format, point-of-care antibody test kits that detect both IgM and IgG antibodies to recombinant viral proteins. The goal is to test at least five (5) different kits including at least two (2) that are manufactured in the USA.

Test procedures. Manufacturers' package inserts or protocols for test performance will be followed. These vary across different test platforms. Persons who perform the tests will not know PCR results or other metadata associated with the human samples when they perform the tests. Tests will be read by two independent readers and recorded. A third reader will be the deciding vote for cases with discordant readings.

Test data. Antibody test results (IgM and IgG) for each different test kit will be entered into a test result form with the participant's unique identifier number (UI). Results will later be merged into a database that contains the UI and metadata such as age, sex, fever, cough, date sample was collected, date of symptom onset, exposure history (travel, household, work). Acceptability of test performance will be judged according to a working target product profile (TPP) appended at the end of this protocol.

Primary objective

1. To assess the sensitivity and specificity of tests for antibody to SARS-CoV-2, the virus that causes COVID-19 disease. Separate criteria will be used to define sensitivity for acute and convalescent samples.

1. Sensitivity for diagnosis of acute cases will be defined as % positivity in samples from symptomatic cases with positive RT-PCR results. .
2. Sensitivity for detecting antibody in convalescent samples expressed as % will be the number of positive antibody tests divided by the number of samples tested from persons with documented past infections (by RT-PCR) who are now at least 2 weeks past resolution of symptoms and currently RT-PCR negative.
3. Sensitivity will also be defined as % agreement with results from a reference antibody test as soon as one is identified.
4. Specificity will be defined as the % of negative control samples (collected prior to 1/1/2020) that have negative antibody test results.

Secondary Objectives

1. To determine relationships between the time after infection or onset of symptoms of COVID-19 and the presence of antibodies to the virus as determined by antibody test kits.
2. To determine the duration of antibody responses following infection.
3. To compare background reactivity (false positive rates) for sera from the USA vs. sera from developing countries in areas where chronic parasitic infections and consumption of bushmeat are common or where people live in close relationship with wildlife that may be a reservoir for zoonotic viruses.
4. To assess test performance characteristics (ease of use).

Benefits to participants. None

Benefits to society. Antibody tests may be useful for diagnosis of infection and for documentation of past infection. Independent test validation studies are critically important. That is because test results from companies may be biased. In addition, companies often do not report on the user friendliness of rapid diagnostics. Antibody tests may be especially valuable for use in low and middle income countries that lack resources for widespread molecular testing for SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* Sera/plasma from patients who have been hospitalized and tested positive for SARS-CoV-2
* Sera/plasma from people who have recovered from COVID-19
* Sera/plasma from from healthy humans and persons with parasitic diseases

Exclusion Criteria:

* Persons under the age of 18

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Sera/plasma from patients in St. Louis, Missouri who have been hospitalized and tested positive for SARS-CoV-2
  * Sera/plasma from people in St. Louis, Missouri who have recovered from COVID-19
  * Sera/plasma from from healthy humans in the US and from rural areas of low and middle income countries
  Note: No voluntary enrolment into this study will be conducted; all testing is to be conducted anonymously.
Sampling Method: Non-Probability Sample
Enrollment: 461 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
Test Sensitivity | 2020
  Test sensitivity relative to RT-PCR for acute samples; sensitivity relative to ELISA for convalescent samples.
Test Specificity | 2020
  Percent positivity with pre-COVID samples

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Bogus J, Gankpala L, Fischer K, Krentel A, Weil GJ, Fischer PU, Kollie K, Bolay FK. Community Attitudes Toward Mass Drug Administration for Control and Elimination of Neglected Tropical Diseases After the 2014 Outbreak of Ebola Virus Disease in Lofa County, Liberia. Am J Trop Med Hyg. 2016 Mar;94(3):497-503. doi: 10.4269/ajtmh.15-0591. Epub 2015 Dec 14. PMID 26666700
- [Background] Chesnais CB, Awaca-Uvon NP, Bolay FK, Boussinesq M, Fischer PU, Gankpala L, Meite A, Missamou F, Pion SD, Weil GJ. A multi-center field study of two point-of-care tests for circulating Wuchereria bancrofti antigenemia in Africa. PLoS Negl Trop Dis. 2017 Sep 11;11(9):e0005703. doi: 10.1371/journal.pntd.0005703. eCollection 2017 Sep. PMID 28892473
- [Background] Corman VM, Landt O, Kaiser M, Molenkamp R, Meijer A, Chu DK, Bleicker T, Brunink S, Schneider J, Schmidt ML, Mulders DG, Haagmans BL, van der Veer B, van den Brink S, Wijsman L, Goderski G, Romette JL, Ellis J, Zambon M, Peiris M, Goossens H, Reusken C, Koopmans MP, Drosten C. Detection of 2019 novel coronavirus (2019-nCoV) by real-time RT-PCR. Euro Surveill. 2020 Jan;25(3):2000045. doi: 10.2807/1560-7917.ES.2020.25.3.2000045. PMID 31992387
- [Background] Li Z, Yi Y, Luo X, Xiong N, Liu Y, Li S, Sun R, Wang Y, Hu B, Chen W, Zhang Y, Wang J, Huang B, Lin Y, Yang J, Cai W, Wang X, Cheng J, Chen Z, Sun K, Pan W, Zhan Z, Chen L, Ye F. Development and clinical application of a rapid IgM-IgG combined antibody test for SARS-CoV-2 infection diagnosis. J Med Virol. 2020 Sep;92(9):1518-1524. doi: 10.1002/jmv.25727. Epub 2020 Apr 13. PMID 32104917
- [Background] Okba NMA, Muller MA, Li W, Wang C, GeurtsvanKessel CH, Corman VM, Lamers MM, Sikkema RS, de Bruin E, Chandler FD, Yazdanpanah Y, Le Hingrat Q, Descamps D, Houhou-Fidouh N, Reusken CBEM, Bosch BJ, Drosten C, Koopmans MPG, Haagmans BL. Severe Acute Respiratory Syndrome Coronavirus 2-Specific Antibody Responses in Coronavirus Disease Patients. Emerg Infect Dis. 2020 Jul;26(7):1478-1488. doi: 10.3201/eid2607.200841. Epub 2020 Jun 21. PMID 32267220
- [Background] Tang YW, Schmitz JE, Persing DH, Stratton CW. Laboratory Diagnosis of COVID-19: Current Issues and Challenges. J Clin Microbiol. 2020 May 26;58(6):e00512-20. doi: 10.1128/JCM.00512-20. Print 2020 May 26. PMID 32245835
- [Background] Weil GJ, Curtis KC, Fakoli L, Fischer K, Gankpala L, Lammie PJ, Majewski AC, Pelletreau S, Won KY, Bolay FK, Fischer PU. Laboratory and field evaluation of a new rapid test for detecting Wuchereria bancrofti antigen in human blood. Am J Trop Med Hyg. 2013 Jul;89(1):11-15. doi: 10.4269/ajtmh.13-0089. Epub 2013 May 20. PMID 23690552
- [Background] Weil GJ, Lammie PJ, Weiss N. The ICT Filariasis Test: A rapid-format antigen test for diagnosis of bancroftian filariasis. Parasitol Today. 1997 Oct;13(10):401-4. doi: 10.1016/s0169-4758(97)01130-7. PMID 15275155